CLINICAL TRIAL: NCT03331315
Title: A Randomized Control Trial Study of the Efficacy of Celecoxib Versus Ketorolac for Perioperative Pain Control
Brief Title: Toradol v. Celecoxib for Postoperative Pain
Acronym: POP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Ulm, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Ulm, MD, Priniciple Investigator, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-02041-FB
Record Dates: First submitted 2015-04-07; First posted 2017-11-06 (Actual); Results first posted 2018-06-04 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Active Comparator): Patients receiving scheduled ketorolac postoperatively
  Interventions: Drug: Ketorolac
- Celecoxib (Experimental): Patients receiving celebrex preoperative and postoperatively for 7 days
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib
  Arms: Celecoxib
Drug: Ketorolac
  Arms: Ketorolac

SUMMARY:
Randomized control trial between ketorolac versus celecoxib for postoperative pain following hysterectomy.

DETAILED DESCRIPTION:
Purpose:

To determine if Celebrex (Celecoxib) is as effective as Toradol (Ketorolac) at controlling postoperative pain when given in addition to standard postoperative pain control regimens.

Rationale:

Toradol (Ketorolac) is currently used by many surgeons as adjuvant therapy in addition to standard narcotics in managing immediate postoperative pain. Toradol (Ketorolac) is a non-steroidal anti-inflammatory drug that acts as a non-selective cyclooxygenase (COX), inhibiting COX-1 and COX-2 isoforms. (Toradol) Ketorolac has been associated with significant complications including postoperative bleeding and acute renal insufficiency. Celebrex (Celecoxib) is a selective COX-2 inhibitor that has been associated with adverse cardiovascular outcomes in patients with pre-existing cardiac disease but not with postoperative bleeding or renal insufficiency. Celebrex (Celecoxib) has also been shown to control postoperative pain but has never been compared to Toradol (Ketorolac).

Population:

Patients undergoing hysterectomy on the gynecology oncology service.

Design:

Randomized control trial.

Procedures:

All patients will receive a standard postoperative pain regimen with oral Tylenol (Acetaminophen), oral Lortab (Hydrocodone/Acetaminophen) as needed, and IV Dilaudid (Hydromorphone) as needed.

Randomization: Each participant will be assigned a number using a random number generator for assignment to one of the two postoperative pain regimens:

Arm 1:

Patients ages 18-65 will receive IV Toradol (Ketorolac) 30mg q6 hrs after their operation for 48 hrs or until hospital discharge if patients are discharged home in less than 48 hours after their operation.

**Patients over age 65 will receive IV Toradol (Ketorolac) 15mg q6hrs instead of 30mg

Arm 2:

Patients who will receive oral Celebrex (Celecoxib) 400mg 1 hour prior to their procedure then 200mg oral twice daily for a total of seven days. Patients discharged prior to 7 days will be given a prescription for Celebrex (Celecoxib) to complete a total of 7 days.

Following surgery all patients will be given a postoperative questionnaire at the day of surgery, which was returned at the two week postoperative visit, examining time until return to ADLs, days of narcotic use, and number of narcotic pills used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hysterectomy

Exclusion Criteria:

* Coronary Artery Disease
* Peptic Ulcer Disease
* Chronic Renal Disease
* Liver disease
* Alcohol Abuse
* Daily narcotic usage
* Narcotic use 24 hours prior to surgery
* Crohn's Disease
* History of myocardial infarction
* History of stroke
* Preoperative hematocrit less than 24
* Asthma
* Ulcerative Colitis
* Diverticulitis
* Aspirin Allergy
* Sulfonamide Allergy
* Pre-operative pain score of greater than 3
* Patients undergoing procedures that may involve bowel resection or bowel reanastomosis.
* Allergy to any non-steroidal anti-inflammatory drug
* Cardiac anomaly or disease
* Congestive Heart Failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Ulm, MD, Principal Investigator — University of Tennessee
Locations (1):
- Methodist Hospital System, Memphis, Tennessee, United States

REFERENCES:
- [Background] Azari L, Santoso JT, Osborne SE. Optimal pain management in total abdominal hysterectomy. Obstet Gynecol Surv. 2013 Mar;68(3):215-27. doi: 10.1097/OGX.0b013e31827f5119. PMID 23945838
- [Background] Blanton E, Lamvu G, Patanwala I, Barron KI, Witzeman K, Tu FF, As-Sanie S. Non-opioid pain management in benign minimally invasive hysterectomy: A systematic review. Am J Obstet Gynecol. 2017 Jun;216(6):557-567. doi: 10.1016/j.ajog.2016.12.175. Epub 2016 Dec 30. PMID 28043841
- [Background] Strom BL, Berlin JA, Kinman JL, Spitz PW, Hennessy S, Feldman H, Kimmel S, Carson JL. Parenteral ketorolac and risk of gastrointestinal and operative site bleeding. A postmarketing surveillance study. JAMA. 1996 Feb 7;275(5):376-82. PMID 8569017
- [Background] Gong L, Thorn CF, Bertagnolli MM, Grosser T, Altman RB, Klein TE. Celecoxib pathways: pharmacokinetics and pharmacodynamics. Pharmacogenet Genomics. 2012 Apr;22(4):310-8. doi: 10.1097/FPC.0b013e32834f94cb. No abstract available. PMID 22336956

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac: Patients receiving scheduled ketorolac postoperatively
  Ketorolac
- Celecoxib: Patients receiving celebrex preoperative and postoperatively for 7 days
  Celecoxib
Period: Overall Study
Arm/Group | Ketorolac | Celecoxib
Started | 88 | 82
Completed | 70 | 68
Not Completed | 18 | 14
Not completed — Physician Decision | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Celecoxib | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11.3) | 55.1 (14.4) | 55.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 31.8 (8.6) | 31.7 (8.1) | 31.7 (8.3)
Surgical Pathology [Count of Participants; unit: Participants]
  Benign | 48 | 53 | 101
  Malignant | 22 | 15 | 37
Procedure [Count of Participants; unit: Participants] — BSO - bilateral salpingo-oophorectomy LND - Lymph Node Dissection Cysto - diagnostic cystoscopy
  Participants
    Robotic Assisted Hysterectomy, +/- BSO, Cysto | 48 | 53 | 101
    Robotic Assisted Hysterectomy, +/- BSO, LND, Cysto | 22 | 15 | 37
Operative Time [Mean (Standard Deviation); unit: Minutes] | 105 (32) | 104 (34) | 104 (33)
Trochar Sites [Mean (Standard Deviation); unit: Trochars] | 4.3 (0.5) | 4.2 (0.4) | 4.2 (0.5)
Preoperative Diagnosis [Count of Participants; unit: Participants]
  Malignancy | 21 | 15 | 36
  Premalignancy | 14 | 15 | 29
  Leiomyoma | 8 | 4 | 12
  Pelvic Pain | 11 | 8 | 19
  Abnormal Uterine Bleeding | 3 | 8 | 11
  Adnexal Mass | 10 | 14 | 24
  Genetic Predisposition to Malignancy | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Average Inpatient Postoperative Pain Score
Description: Pain measured using the Visual Analog Scale, no pain (0-0.4 cm), mild pain(0.5-4.4 cm), moderate pain (4.5-7.4 cm), and severe pain (7.5-10.0 cm). Subscale scoring was not used in analysis but provided as reference for patient and nursing staff.
Time Frame: 48 hrs following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
units on a scale | 2.7 (1.9) | 2.4 (1.6)

2. Secondary Outcome: Average Inpatient Hydromorphone Use
Description: Average inpatient hydromorphone use measured in milligrams
Time Frame: 48 hrs following surgery
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Milligrams | 0.7 (1.0) | 0.8 (1.0)

3. Secondary Outcome: Average Inpatient Ondansetron Use
Description: Average inpatient ondansetron use measured in milligrams
Time Frame: 48 hrs following surgery
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Milligrams | 1.5 (1.9) | 1.3 (2.2)

4. Secondary Outcome: Total Hospital Stay
Description: Total hospital stay from time fo admission to time of discharge measured in hours
Time Frame: Following surgery
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Hours | 11.6 (8.1) | 11.9 (7.6)

5. Secondary Outcome: Number of Participants With Perioperative Complications
Description: Perioperative Complications measured intraoperatively and postoperatively by type
Time Frame: During and after surgery
Measure: Number; unit: Patients
Groups:
- Ketorolac; Celecoxib: Participants
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Patients | 5 | 6

6. Secondary Outcome: Return to Activities of Daily Living
Description: Average number of days required for complete return to independent activities of daily living
Time Frame: 2 weeks after discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Days | 2.4 (0.8) | 2.2 (0.9)

7. Secondary Outcome: Days of Oral Narcotic Use After Discharge
Description: Measured using postoperative questionnaire
Time Frame: 2 weeks after discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Days | 5.7 (2.8) | 3.8 (2.6)

8. Secondary Outcome: Number of Oral Narcotic Pills Used After Discharge
Description: Number of oral narcotic pills used after discharge until 2 week postoperative visit.
Time Frame: 2 weeks after discharge
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Ketorolac | Celecoxib
Number analyzed (Participants) | 70 | 68
Pills | 8.1 (4.0) | 6.0 (3.6)

ADVERSE EVENTS:
Arm/Group | Ketorolac | Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 1/70 | 2/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=70) | Celecoxib (N=68)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Transient acute kidney injury, resolved with IV hydration
Intraoperative Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Estimated Blood Loss >150cc

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No